CLINICAL TRIAL: NCT06485778
Title: Phase 2 Single Arm Trial of Adjuvant Nodal Irradiation Alone in Post Operative Oral Tongue Squamous Cell Carcinoma
Brief Title: A Study of Radiation Therapy After Surgery in People With Oral Tongue Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-167
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Oral Tongue Squamous Cell Carcinoma
Keywords: pT1-2,pN0-2b; intensity modulated radiation therapy (IMRT); 24-167
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Phase 2 single arm trial enrolling post operative oral tongue squamous cell carcinoma patients with pT1-2N0-N2b.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy (Experimental): These patients will then receive bilateral cervical nodal irradiation with the primary post operative site excluded (30 fractions). They will be monitored for both physician reported toxicities.
  Interventions: Radiation: Photon intensity modulated radiation therapy (IMRT); Other: Life questionnaire's

INTERVENTIONS:
Radiation: Photon intensity modulated radiation therapy (IMRT) — Patients will receive bilateral cervical nodal irradiation with the primary post operative site excluded (30 fractions).
Other: Life questionnaire's — EORTC QLQ C30/HN 35 and MDADI

SUMMARY:
This study will test whether limiting standard photon intensity modulated radiation therapy (IMRT) to exclude the oral tongue surgical site can decrease the risk of side effects caused by oral radiation. The researchers will also find out if this approach affects the rate of disease coming back after treatment (recurrence), and will measure participants' quality of life by having them complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Surgical resection of all gross disease without evidence of residual loco-regional disease on simulation PET/CT.
* pT1-2, or pT3 by DOI, pN0-2b Squamous Cell Carcinoma of the Oral Tongue confirmed on final surgical pathology. Patients must have:

  * at least two of the following pathologic risk features

    * LVI
    * DOI ≥ 4mm and ≤ 10mm OR
  * 1 or 2 pathologically positive nodes N1 to low volume N2b. OR DOI >10 mm OR
  * <=cT3N2b who undergo induction with near pCR (<5% viable) or pCR at primary site
* Primary specimen surgical margins ≥3 mm (if <WPOI 5, margin can be >= 2.2mm)
* Signed informed consent form by the participant or their legally authorized representative (LAR)

Exclusion Criteria:

* N2c/N3 nodal disease
* pT3 by size
* >2 pathologically positive nodes
* Primary specimen surgical margin < 3 mm
* Extensive Perineural Invasion (PNI); non-extensive PNI is permitted.
* Extra-capsular extension in any pathologically positive lymph node
* Prior or simultaneous invasive malignancy that, in the opinion of the PI, represents a competing risk of death equivalent to the patient's oral tongue squamous cell carcinoma.
* Auto-immune conditions that would otherwise preclude radiation in the opinion of the PI (e.g. Scleroderma).
* Lack of ability to understand and willingness to sign a written informed consent and complete questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Acute Grade ≥3 Oral Mucositis | within 120 days of radiation completion
  This is defined by CTCAE v 5.0 criteria

SECONDARY OUTCOMES:
Cumulative Incidence of Local Failure | 2 years
  will be defined as any local failure in the oral tongue/FOM/BOT that is subsequently proven by biopsy during protocol-mandated follow-up. Competing risks will be distant or regional failure without local failure or death without progression. This will be calculated from the start of radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Sean McBride, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm